CLINICAL TRIAL: NCT06811350
Title: Quality Improvement Initiative for Enhancing Early Mobilization in Intracerebral Hemorrhage Patients: Pre-Post Implementation of a Structured Clinical Pathway
Brief Title: Quality Improvement Initiative for Enhancing Early Mobilization in Intracerebral Hemorrhage Patients
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202410128RINB
Record Dates: First submitted 2025-01-13; First posted 2025-02-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-11

CONDITIONS: Primary Intracerebral Hemorrhage; Early Mobilization
Keywords: Intracerebral hemorrhage; Early mobilization; Stroke unit; Clinical pathway
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pre-implementation cohort: Patients received conventional care without a structured mobility pathway, with mobilization decisions made at the discretion of the attending physician and rehabilitation team.
  Interventions: Procedure: post-implementation cohort

INTERVENTIONS:
Procedure: post-implementation cohort — Patients recieved a structured early mobilization pathway was introduced. The pathway included standardized assessments for patient stability and phased rehabilitation, progressing from passive to active mobilization.

SUMMARY:
Primary intracerebral hemorrhage (ICH) is a severe and life-threatening condition with a high mortality rate, reaching up to 50% within the first month. Survivors are often at risk of long-term disability due to the extensive brain damage caused by the hemorrhage. Unlike ischemic stroke patients, ICH patients are typically younger, face longer hospital stays, and are more likely to experience acute complications. Modern treatment approaches have shifted from focusing solely on reducing mortality to minimizing disability and enhancing functional outcomes through early rehabilitation. However, the optimal timing and intensity of early mobilization remain unclear, especially for patients with severe ICH, where medical stability is a major concern. Delays in initiating rehabilitation may limit neuroplasticity and hinder recovery, prompting the need for a structured, multidisciplinary approach to early mobilization in ICH patients.

Objective : This quality improvement (QI) initiative aimed to enhance early mobilization in ICH patients by implementing a structured clinical pathway in an academic stroke center. The goal was to integrate evidence-based early mobilization pathways to improve patient mobility outcomes while ensuring safety through standardized assessments of cardiovascular, respiratory, and neurological stability.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary ICH
* ICH score from 0 to 4
* Patients In line with the stroke center's standard criteria for early rehabilitation

Exclusion Criteria:

* Patients with traumatic brain injury, hemorrhagic transformation of ischemic stroke, or hemorrhage related to underlying malignancy
* Patients placed in palliative care or those who died before initial hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary intracerebral hemorrhage (ICH), a severe and life-threatening condition characterized by bleeding within the brain, carries a high mortality rate of up to 50% within the first month. Survivors of ICH are at significant risk of long-term disability due to the extensive damage caused by the hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 198 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-11-12 (Estimated)

PRIMARY OUTCOMES:
Modified ICU mobility scale | through study completion, an average of 12 weeks
  The Modified ICU Mobility Scale is used to assess the level of mobility in ICU patients, with scores ranging from 0 to 10. A higher score indicates better mobility, where 0 represents no mobility (lying in bed, passive movements only), and 10 indicates independent ambulation without assistance.

SECONDARY OUTCOMES:
the time to first mobilization | Through study completion, an average of 12 weeks
  The time to first mobilization (in hours or days) will be assessed from hospital admission to the first documented mobilization event, measured through study completion, with an average follow-up period of 12 weeks.
National Institutes of Health Stroke Scale (NIHSS) score | through study completion, an average of 12 weeks
  The National Institutes of Health Stroke Scale (NIHSS) is used to assess stroke severity, with scores ranging from 0 to 42. A higher score indicates a worse neurological impairment, where 0 represents no stroke symptoms, and higher scores reflect increasing severity of stroke-related deficits.
Modified Rankin Scale (mRS) | through study completion, an average of 12 weeks
  The Modified Rankin Scale (mRS) is used to assess functional outcomes, with scores ranging from 0 to 6. A higher score indicates a worse outcome, where 0 represents no symptoms, and 6 indicates death.
Duration of ICU and hospital stays | Through study completion, an average of 12 weeks
  The duration of ICU stay (in days) and total hospital stay (in days) will be assessed through study completion, with an average follow-up period of 12 weeks.
ability to ambulate upon discharge | through study completion, an average of 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Tiapei, Taiwan